CLINICAL TRIAL: NCT06149520
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Study to Assess the Efficacy and Safety of BAY 3018250 in Patients With Symptomatic Proximal Deep Vein Thrombosis
Brief Title: A Study to Learn More About How Well BAY3018250 Works and How Safe it is for People With Proximal Deep Vein Thrombosis
Acronym: SIRIUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22138; 2023-503315-15-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-11-15; First posted 2023-11-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Thrombolysis; Symptomatic Proximal Deep Vein Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- BAY3018250 Dose 1 (Experimental): Participants will receive BAY3018250 Dose 1.
  Interventions: Drug: BAY3018250
- BAY3018250 Dose 2 (Experimental): Participants will receive BAY3018250 Dose 2.
  Interventions: Drug: BAY3018250
- Placebo to BAY3018250 (Placebo Comparator): Participants will receive placebo to BAY3018250.
  Interventions: Drug: Placebo to BAY3018250

INTERVENTIONS:
Drug: BAY3018250 — Dose 1 or dose 2 of BAY3018250
  Arms: BAY3018250 Dose 1; BAY3018250 Dose 2
Drug: Placebo to BAY3018250 — Matching placebo to BAY3018250
  Arms: Placebo to BAY3018250

SUMMARY:
Researchers are looking for a better way to treat people who have deep vein thrombosis (DVT).

DVT is a condition that occurs when a blood clot forms in a deep vein in the leg. DVT is called 'proximal' when the clot is formed in the veins of the hip, thigh, and knee. DVT can cause serious health problems. The blood clots in the veins can break loose and can then travel through the bloodstream and get stuck in the lungs, blocking blood flow to the lungs. Symptoms of DVT include swelling, pain, and tenderness in the affected leg, as well as redness and warmth in the area. Currently, DVT is usually treated using blood thinners to prevent the clot from getting bigger or breaking off and traveling to the lungs. However, blood thinners may not be able to remove a blood clot quickly and may not be suitable for everyone who has DVT.

BAY3018250 is a drug that works by dissolving blood clots. In this study, researchers will compare BAY3018250 with placebo to learn how well it works and how safe it is in participants with proximal DVT. A placebo looks like the study drug but does not have any medicine in it. Using a placebo helps researchers to confirm that the results observed during the study were caused by the study drug and not by other factors.

The main purposes of this study are to learn:

* How well BAY3018250 works in dissolving blood clots in participants with proximal DVT and
* How safe is BAY3018250 as a treatment for participants with proximal DVT?

For this, the researchers will use ultrasound tests to measure blood clots in participants before and at various times after study treatment. They call these measurements a clot burden score. They will compare the clot burden score before and after treatment and will calculate a complex measure called AUC. This tells researchers how the clots have changed over time.

And researchers will collect the number of bleeding events that require medical attention.

The study participants will be randomly (by chance) assigned to one of 3 treatment groups. Dependent on the group, they will receive a single dose of high dose or low dose of BAY3018250 or placebo.

Researchers will closely monitor participants for 90 days after receiving the study treatment.

During the study, the doctors and their study team will:

* take blood samples
* do physical examinations
* examine heart health using electrocardiogram (ECG)
* check vital signs such as blood pressure, heart rate
* undergo ultrasound tests to measure the blood clots
* ask the participants questions about how they are feeling and what adverse events they are having.

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events, irrespective if they think it is related or not to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Male and female (if postmenopausal or hysterectomized) aged 18 years or older
* Acute symptomatic proximal deep vein thrombosis (DVT) documented by compression ultrasound (CUS) and all of the following:

  * duration of symptoms 14 days or less
  * Proximal DVT involving at least 1 of the following proximal veins: the popliteal vein, the femoral vein, the common femoral vein and the external iliac vein
  * adequate visualization of the most proximal end of the thrombus
  * receiving therapeutic dose anticoagulation with low molecular weight heparins (LMWHs) and/or direct oral anticoagulants (DOACs) according to the respective product labels
* Measured body weight within 50 to 130 kg
* Signed informed consent

Exclusion Criteria:

* Acute symptomatic pulmonary embolism (PE) requiring systemic or catheter-directed thrombolytic therapy, catheter-directed mechanical thrombectomy, or surgical embolectomy
* Active bleeding or high risk for bleeding (at the discretion of the investigator)
* Recent (<3 months) ischemic stroke, myocardial infarction, intracranial hemorrhage, or major surgery or severe trauma (at the discretion of the investigator)
* Active cancer, i.e., locally active, regionally invasive or metastatic and/or anticancer therapy within the last 6 months, except basal cell or squamous cell carcinoma
* Therapeutic-dose anticoagulants for > 72 hours before randomization, or current use of vitamin K antagonists
* Planned or current use of the following medications:

  * Any antiplatelet therapy, except acetylsalicylic acid (ASA) ≤100 mg/day
  * Antifibrinolytic drugs
  * Therapeutic antibodies
* Male participants with women of childbearing potential (WOCBP) partners unwilling to use highly effective contraception from start of study intervention until end of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
AUCn(6h-30d) of the ratio to baseline of clot burden, as assessed by repeated quantitative ultrasound | at 6 hours, 24 hours, Day 7, Day 30
  Area under the curve (AUC) with respect to the measurement time points at 6 hours, 24 hours, 7 days and 30 days of the ratio to baseline of clot burden
Number of participants with composite of major and clinically relevant non-major (CRNM) bleeding events (ISTH definition) | up to Day 15
  The classify of bleeding events use the International Society on Thrombosis and Haemostasis (ISTH) definitions.

SECONDARY OUTCOMES:
Ratio to baseline of clot burden, as assessed by quantitative ultrasound | at 6 hours, 24 hours, Day 7, Day 30 and Day 90
Change from baseline in leg pain severity | at 6 hours, 24 hours, Day 7, Day 30 and Day 90
  Likert pain scale is used as a quantitative measure of patient reported pain based on the participant´s judgement. The scale ranges from 0 (no pain) to 10 (worst imaginable pain).
Change from baseline in PVFS scale | at Day 7, Day 30 and Day 90
  PVFS stands for post venous thromboembolism functional status. PVFS scale is ordinal, has 6 steps ranging from 0 (no symptoms) to 5 (death), with higher scores being worse and covers the entire range of functional outcomes by focusing on limitations in usual duties/activities either at home or at work/study, as well as changes in lifestyle.
Number of participants with recurrent venous thromboembolism | up to Day 90

CONTACTS AND LOCATIONS:
Locations (68):
- Belgium (7):
  - Universiteit Ziekenhuis Antwerpen | Thoraxheelkunde Afdeling, Antwerp
  - Imelda - Vascular Surgery Dept, Bonheiden
  - Ziekenhuis Oost-Limburg | Genk, Sint-Jan campus - Thoracic Vascular Surgery Department, Genk
  - UZ Gent, Ghent
  - AZ Groeninge - Campus Kennedylaan, Kortrijk
  - Katholieke Universiteit Leuven (KU Leuven) - Center for Molecular and Vascular Biology (CMVB), Leuven
  - AZ Sint-Maarten, Mechelen
- Bulgaria (6):
  - University Multiprofile Hospital For Active Treatment Kanev AD, Rousse
  - Specialized Hospital For Active Cardiology Treatment Medica Kor EAD, Rousse
  - University Multiprofile Hospital For Active Treatment 'Alexandrovska' EAD, Sofia
  - University Multiprofile Hospital for Active Treatment 'Sveta Ekaterina' EAD, Sofia, Sofia
  - Medical Institute Ministry of Interior, Sofia
  - Multiprofile Hospital for Active Treatment Dr. Stefan Cherkezov | Base 1 - Cardiology Department, Veliko Tarnovo
- McGill University Health Centre - Glen Site, Montreal, Quebec, Canada
- Czechia (6):
  - Vojenská nemocnice Brno - Interní oddelení, pododbor kardiologie, Brno
  - Interni oddeleni, Krnovska nemocnice, Sdruzene zdravotnicke zarizeni Krnov, prispevkova organizace, Krnov
  - Kardiologicka klinika, Fakultni nemocnice Kralovske Vinohrady, Prague
  - Všeobecná fakultní nemocnice v Praze - II. interní klinika - klinika kardiologie a angiologie, AJIP, Prague
  - Nemocnice Roudnice nad Labem - interni oddeleni, Roudnice nad Labem
  - Interni a kardiologicka ambulance, Nemocnice Znojmo, prispevkova organizace, Znojmo
- France (10):
  - Centre Hospitalier Universitaire Amiens Picardie Site Sud, Amiens Cedex1
  - Centre Hospitalier Regional Universitaire (CHRU) Brest - Hopital de la Cavale Blanche, Brest
  - Centre Hospitalier Universitaire de Clermont Ferrand - Gabriel Montpied, Clermont-Ferrand
  - Hôpital Louis Mourier - Colombes Cedex, Colombes
  - Centre Hospitalier Universitaire Grenoble Alpes (CHU Grenoble Alpes) - Hopital Albert Michallon, La Tronche
  - AP-HP Hopital Europeen Georges-Pompidou (HEGP) - Service de medecine vasculaire, Paris
  - Centre Hospitalier Universitaire (CHU) de Saint-Etienne - Hopital Nord, Saint-Etienne
  - Hopitaux Universitaires de Strasbourg - Le Nouvel Hopital Civil (NHC), Strasbourg
  - Hôpital Sainte Musse, Toulon
  - Centre Hospitalier Universitaire (CHU) de Toulouse - Hopital de Rangueil - Service de medecine vasculaire, Toulouse
- Germany (4):
  - UNIVERSITAETSKLINIKUM FREIBURG - Universitaets-Herzzentrum Bad Krozingen | Klinik für Kardiologie und Angiologie, Bad Krozingen
  - Universitaetsklinikum Carl Gustav Carus an der Technischen Universitaet Dresden | Medizinische Klinik I - FB Haemostaseologie, Dresden
  - LMU Klinikum Campus Innenstadt | Medizinische Klinik und Poliklinik IV | FB Angiologie, München
  - Universitaetsklinikum Muenster | Klinik fuer Kardiologie I Sektion Angiologie, Münster
- Greece (5):
  - General Hospital Of Athens G Gennimatas- Department of Vascular Surgery, Athens
  - University General Hospital Attikon - 1st Department of Vascular surgery University of Athens, Athens
  - General Hospital Of Thessaloniki Papageorgiou- 1st Department of Surgery, Efkarpia
  - University General Hospital Of Ioannina- Department of Surgery, Vascular Unit Faculty, Ioannina
  - General University Hospital Of Patras- Department of Vascular Surgery, Pátrai
- Hungary (6):
  - Bekes Varmegyei Kozponti Korhaz - Dr. Rethy Pal Tagkorhaz, Békéscsaba
  - Semmelweis Egyetem - Belgyógyászati és Hematológiai Klinika, Kardiológia, Budapest
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz - Általános Belgyógyászati Osztály, Kaposvár
  - Kistarcsai Flor Ferenc Korház - II. Belgyógyászat - Angiológia, Kistarcsa
  - Szegedi Tudományegyetem, Szent-Györgyi Albert Klinikai Központ - Belgyógyászati Klinika, Szeged
  - Fejer Varmegyei Szent Gyorgy Egyetemi Oktato Korhaz - II. Belgyogyaszat, Székesfehérvár
- Italy (8):
  - Azienda Ospedaliero-Universitaria Di Bologna IRCCS_Policlinico Sant'Orsola - Angiologia e Malattie della Coagulazione, Bologna
  - Azienda Unita Locale Socio Sanitaria 2 Marca Trevigiana | Castelfranco Veneto Hospital - Angiologia Department, Castelfranco Veneto
  - Azienda Ospedale-Università di Padova - Medicina Generale ad indirizzo trombotico-emorragico, Padua
  - Azienda Unita Sanitaria Locale di Reggio Emilia | Arcispedale Santa Maria Nuova - Cardiovascular Medicine, Reggio Emilia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOSD Malattie Emorragiche e Trombotiche, Roma
  - Humanitas Mirasole S.p.A. - Centro Trombosi e Malattie Emorragiche, Rozzano
  - AULSS N. 2 Marca Trevigiana_Ospedale di Treviso - UOC Pronto Soccorso, Treviso
  - ASST dei Sette Laghi | Ospedale Di Circolo e Fondazione Macchi Di Varese - Centro Trombosi ed Emostasi, Varese
- Netherlands (3):
  - Albert Schweitzer Hospital | Internal Medicine - Hematology Department, Dordrecht
  - Zuyderland Medical Centre | Internal Medicine Department, Geleen
  - Leids Universitair Medisch Centrum (LUMC) (Leiden University Medical Center), Leiden
- Slovakia (5):
  - Penta Hospitals | Zeleznicna Nemocnica Kosice - Angiologicka ambulancia, Košice
  - Kardiocentrum AGEL a.s. - Angiologické oddelenie, Košice
  - Nemocnicná a.s. - Interné oddelenie, Malacky
  - Penta Hospitals | Hospital and Polyclinic Spisska Nova Ves - Internal Medicine Department, Spišská Nová Ves
  - Hospitale, s.r.o. - Interné oddelenie, Šahy
- Spain (2):
  - Hospital Universitario Infanta Sofia | Medicina Interna, San Sebastián de los Reyes, Madrid
  - Hospital Universitari De Girona Doctor Josep Trueta | Medicina Interna, Girona
- Turkey (Türkiye) (5):
  - Ankara Bilkent Sehir Hastanesi, Bilkent Ankara
  - Istanbul Universitesi Cerrahpasa-Cerrahpasa Tip Fakultesi, Istanbul
  - Saglik Bilimleri Üniversitesi Dr. Siyami Ersek Gögüs Kalp ve Damar Cerrahisi Egitim Ve Arastirma Hastanesi, Istanbul
  - Izmir Sehir Hastanesi, Izmir
  - Erciyes Universitesi Tip Fakultesi, Kayseri

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — https://clinicaltrials.bayer.com/study/22138